CLINICAL TRIAL: NCT07339943
Title: Micro-ultrasound-Guided Focal Laser Ablation (MicroUSgFLA) Treatment for Management of Intermediate-Risk Prostate Cancer: Evaluation of Safety and Effectiveness
Brief Title: Micro-ultrasound-Guided Focal Laser Ablation for Intermediate-Risk Prostate Cancer: Safety & Effectiveness
Acronym: MicroUSgFLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Exact Imaging (Industry); Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-6189
Record Dates: First submitted 2025-09-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Adenocarcinoma); Low and Intermediate Risk Prostate Cancer
Keywords: Micro-Ultrasound Guided Focal Laser Ablation; Focal Therapy; Focal Laser Ablation; Minimally Invasive Treatment; Laser Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Longitudinal Studies

STUDY DESIGN:
Intervention Model Description: 6 Month, Prospective, Interventional, Open-label Single-Arm Effectiveness Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Prospective Clinical Trial (Experimental): This is a single arm study where patients with intermediate risk MR visible locally confined prostate cancer will be treated with Micro-Ultrasound Guided Focal Laser Ablation. Following treatment, the patients will be assessed by MRI and Biopsy at 6 months with PSA.
  Interventions: Procedure: 6 month, prospective, interventional single-arm safety and effectiveness study; Device: The TRANBERG|CLS Thermal therapy

INTERVENTIONS:
Procedure: 6 month, prospective, interventional single-arm safety and effectiveness study — x
  Other Names: MicroUSgFLA treatment; Focal Laser Ablation treatment; Minimally invasive treatments for prostate cancer
Device: The TRANBERG|CLS Thermal therapy — Micro Ultrasound Guided Focal Laser Ablation of Prostate Cancer by The Diode Laser System - The TRANBERGCLS|Thermal Therapy
  Other Names: ExactVu Micro-Ultrasound System

SUMMARY:
This clinical research study is intended to show that Micro-Ultrasound Guided Focal Laser Ablation (MicroUSgFLA) is a safe procedure that can significantly postpone or eliminate the need for patients with intermediate-Risk prostate cancer (PCa) to undergo a definitive treatment (i.e., Radical Prostatectomy or Radiation Therapy) for their disease.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men, and a large proportion of these diagnoses are of the low or intermediate risk type that are amenable to a minimally invasive approach to treatment such as Focal Therapy. If successful, this study will show that trans-perineal interstitial laser focal therapy of the prostate could be offered over a wider community setting than only at a major hospital as an Magnetic Resonance Imaging (MRI), to confidently locate the Index Lesion would not be required because MicroUS is showing the same potential to visualize the lesion. MicroUS-guided focal laser ablation would be a simpler treatment than the complexity required under MRI, it could be offered in communities that might not have local access to MRI facilities and could be offered to individuals who are contra-indicated for MRI for such reasons as having metallic implants or severe claustrophobia.

ELIGIBILITY:
Inclusion Criteria:

* Men 40-80 years of age.
* Histologically-proven intermediate-risk PCa (Gleason score 7, primary grade ≤ 4).
* PCa clinical stage T1c or T2.
* MRI/MicroUS site suspicious for cancer or cancer mapped to one prostate lobe.
* Maximum dimension of MRI/MicroUS visible tumour ≤15mm.
* Suspicious site on Prostate MRI/MicroUS must coincide with sector positive for cancer on biopsy.
* Prostate specific antigen (PSA) level < 15 ng/mL.
* IPSS, ICIQ-UI-SF, IIEF-15 questionnaires completed prior to the procedure.
* Life expectancy of greater than 10 years, based on co-morbidity not related to PCa.

Exclusion Criteria:

* Maximum dimension of MRI/MicroUS visible tumour > 15 mm.
* Patients medically unfit for focal therapy of the prostate.
* Patients who are unwilling or unable to give informed consent.
* Patients who have received androgen suppression therapy.
* Patients who have received or are receiving chemotherapy for prostate carcinoma.
* Patients previously treated with surgery to the prostate (traditional, endoscopic or minimally invasive) including HIFU, TUNA, RITA, microwave, cryotherapy or any curative treatment.
* Patients who have undergone radiation therapy for PCa or to the pelvis.
* Any condition or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies).
* Patients with a history of non-compliance with medical therapy and/or medical recommendations.
* Patients who are unwilling or unable to complete the patient self-assessment questionnaires.
* Chronic or acute prostatitis, neurogenic bladder, urinary tract infection, sphincter abnormalities, or any other symptom that prevents normal micturition.
* Patients who have participated in a clinical study and/or received treatment with an investigational treatment and/or product within the past 90 days.
* Patients with contraindication to MRI (i.e. pacemaker, hip prosthesis, severe claustrophobia, brain aneurysm clip, allergy to MRI contrast agent)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer
Enrollment: 7 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: | From enrollment to the end of treatment at 6 months.
  Number of Participants With Procedure-Related Adverse Events Time Frame: Up to 6 months after procedure Outcome Type: Safety
  Measure Description:
  Number and severity of procedure-related adverse events (AEs), graded according to CTCAE v5.0, to evaluate the safety profile of focal Micro-Ultrasound-Guided Focal Laser Ablation (MicroUS-gFLA) in patients with organ-confined intermediate-risk prostate cancer.
  Unit of Measure: Number of participants
Primary Outcome 2: Technical Success Rate of MicroUS-gFLA | From enrollment to the end of treatment at 6 months
  Primary Outcome 2: Technical Success Rate of MicroUS-gFLA
  Time Frame: At completion of procedure; confirmed during follow-up up to 6 months Outcome Type: Feasibility
  Measure Description:
  Proportion of procedures achieving technical success, defined as: successful visualization and MicroUS-guided trocar insertion into the target lesion, and completion of focal laser ablation exactly as planned, as confirmed by intra-procedural imaging and follow-up mpMRI and/or biopsy. Unit of Measure: Percentage of procedures

SECONDARY OUTCOMES:
Secondary Outcome 1 - Change in PSA Level From Baseline | From enrollment to the end of treatment at 6 months.
  Secondary Outcome 1 - Change in PSA Level From Baseline
  Time Frame: Baseline to 6 months Outcome Type: Efficacy
  Measure Description:
  Change in serum prostate-specific antigen (PSA) level from baseline prior to ablation to 6-month follow-up.
  Unit of Measure: Change in PSA (ng/mL)
Secondary Outcome 2: Change in Urinary Function (IPSS Score) | From enrollment to the end of the treatment at 6 months
  Secondary Outcome 2: Change in Urinary Function (IPSS Score)
  Time Frame: Baseline, 3 months, and 6 months Outcome Type: Functional
  Measure Description:
  Change in urinary function measured using the International Prostate Symptom Score (IPSS).
  Unit of Measure: Change in score (IPSS scale)
Secondary Outcome 3: Change in Erectile Function (IIEF-15 Score) | From enrollment to the end of treatment at 6 months
  Secondary Outcome 3: Change in Erectile Function (IIEF-15 Score)
  Time Frame: Baseline, 3 months, and 6 months Outcome Type: Functional
  Measure Description:
  Change in erectile function measured using the International Index of Erectile Function-15 (IIEF-15) questionnaire.
  Unit of Measure: Change in score (IIEF-15 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeet Ghai, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that relate to the results reported in the primary publication (e.g., baseline demographics, imaging findings, treatment parameters, outcomes, and adverse events).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of the primary results for up to 5 years thereafter.
Access Criteria: Data will be available to investigators with methodologically sound research proposals for use in projects related to prostate imaging, focal therapy, or outcomes research. All requestors will be required to sign a data use agreement to ensure participant confidentiality.
  Data requests should be submitted to the study principal investigator. Approved proposals will be granted access via a secure institutional data-sharing platform.

REFERENCES:
- [Background] Thompson IM, Pauler DK, Goodman PJ, Tangen CM, Lucia MS, Parnes HL, Minasian LM, Ford LG, Lippman SM, Crawford ED, Crowley JJ, Coltman CA Jr. Prevalence of prostate cancer among men with a prostate-specific antigen level < or =4.0 ng per milliliter. N Engl J Med. 2004 May 27;350(22):2239-46. doi: 10.1056/NEJMoa031918. PMID 15163773
- [Background] Thompson IM, Goodman PJ, Tangen CM, Lucia MS, Miller GJ, Ford LG, Lieber MM, Cespedes RD, Atkins JN, Lippman SM, Carlin SM, Ryan A, Szczepanek CM, Crowley JJ, Coltman CA Jr. The influence of finasteride on the development of prostate cancer. N Engl J Med. 2003 Jul 17;349(3):215-24. doi: 10.1056/NEJMoa030660. Epub 2003 Jun 24. PMID 12824459
- [Background] Wheeler WE, Scott-Conner CE, Stone RA. Flexible sigmoidoscopy as a screening procedure for asymptomatic colorectal carcinoma in patients with inguinal hernia. South Med J. 1985 Dec;78(12):1417-20. doi: 10.1097/00007611-198512000-00005. PMID 4071166
- [Background] Lindner U, Lawrentschuk N, Weersink RA, Davidson SR, Raz O, Hlasny E, Langer DL, Gertner MR, Van der Kwast T, Haider MA, Trachtenberg J. Focal laser ablation for prostate cancer followed by radical prostatectomy: validation of focal therapy and imaging accuracy. Eur Urol. 2010 Jun;57(6):1111-4. doi: 10.1016/j.eururo.2010.03.008. Epub 2010 Mar 12. PMID 20346578
- [Background] Lindner U, Weersink RA, Haider MA, Gertner MR, Davidson SR, Atri M, Wilson BC, Fenster A, Trachtenberg J. Image guided photothermal focal therapy for localized prostate cancer: phase I trial. J Urol. 2009 Oct;182(4):1371-7. doi: 10.1016/j.juro.2009.06.035. Epub 2009 Aug 14. PMID 19683262
- [Background] Peters RD, Chan E, Trachtenberg J, Jothy S, Kapusta L, Kucharczyk W, Henkelman RM. Magnetic resonance thermometry for predicting thermal damage: an application of interstitial laser coagulation in an in vivo canine prostate model. Magn Reson Med. 2000 Dec;44(6):873-83. doi: 10.1002/1522-2594(200012)44:63.0.co;2-x. PMID 11108624
- [Background] Guillaumier S, Peters M, Arya M, Afzal N, Charman S, Dudderidge T, Hosking-Jervis F, Hindley RG, Lewi H, McCartan N, Moore CM, Nigam R, Ogden C, Persad R, Shah K, van der Meulen J, Virdi J, Winkler M, Emberton M, Ahmed HU. A Multicentre Study of 5-year Outcomes Following Focal Therapy in Treating Clinically Significant Nonmetastatic Prostate Cancer. Eur Urol. 2018 Oct;74(4):422-429. doi: 10.1016/j.eururo.2018.06.006. Epub 2018 Jun 28. PMID 29960750
- [Background] Alibhai SM, Naglie G, Nam R, Trachtenberg J, Krahn MD. Do older men benefit from curative therapy of localized prostate cancer? J Clin Oncol. 2003 Sep 1;21(17):3318-27. doi: 10.1200/JCO.2003.09.034. PMID 12947068
- [Background] Reddy D, Bedi N, Dudderidge T. Focal therapy, time to join the multi-disciplinary team discussion? Transl Androl Urol. 2020 Jun;9(3):1526-1534. doi: 10.21037/tau.2019.09.30. PMID 32676440
- [Background] Langer DL, van der Kwast TH, Evans AJ, Sun L, Yaffe MJ, Trachtenberg J, Haider MA. Intermixed normal tissue within prostate cancer: effect on MR imaging measurements of apparent diffusion coefficient and T2--sparse versus dense cancers. Radiology. 2008 Dec;249(3):900-8. doi: 10.1148/radiol.2493080236. PMID 19011187
- [Background] Eure G, Fanney D, Lin J, Wodlinger B, Ghai S. Comparison of conventional transrectal ultrasound, magnetic resonance imaging, and micro-ultrasound for visualizing prostate cancer in an active surveillance population: A feasibility study. Can Urol Assoc J. 2019 Mar;13(3):E70-E77. doi: 10.5489/cuaj.5361. Epub 2018 Aug 30. PMID 30169149
- [Background] Weinreb JC, Barentsz JO, Choyke PL, Cornud F, Haider MA, Macura KJ, Margolis D, Schnall MD, Shtern F, Tempany CM, Thoeny HC, Verma S. PI-RADS Prostate Imaging - Reporting and Data System: 2015, Version 2. Eur Urol. 2016 Jan;69(1):16-40. doi: 10.1016/j.eururo.2015.08.052. Epub 2015 Oct 1. PMID 26427566
- [Background] Ghai S, Eure G, Fradet V, Hyndman ME, McGrath T, Wodlinger B, Pavlovich CP. Assessing Cancer Risk on Novel 29 MHz Micro-Ultrasound Images of the Prostate: Creation of the Micro-Ultrasound Protocol for Prostate Risk Identification. J Urol. 2016 Aug;196(2):562-9. doi: 10.1016/j.juro.2015.12.093. Epub 2016 Jan 12. PMID 26791931
- [Background] Klotz L, Lughezzani G, Maffei D, Sanchez A, Pereira JG, Staerman F, Cash H, Luger F, Lopez L, Sanchez-Salas R, Abouassaly R, Shore ND, Eure G, Paciotti M, Astobieta A, Wiemer L, Hofbauer S, Heckmann R, Gusenleitner A, Kaar J, Mayr C, Loidl W, Rouffilange J, Gaston R, Cathelineau X, Klein E. Comparison of micro-ultrasound and multiparametric magnetic resonance imaging for prostate cancer: A multicenter, prospective analysis. Can Urol Assoc J. 2021 Jan;15(1):E11-E16. doi: 10.5489/cuaj.6712. PMID 32701437
- [Background] Johansson JE, Andren O, Andersson SO, Dickman PW, Holmberg L, Magnuson A, Adami HO. Natural history of early, localized prostate cancer. JAMA. 2004 Jun 9;291(22):2713-9. doi: 10.1001/jama.291.22.2713. PMID 15187052
- [Background] McLeod DG, Iversen P, See WA, Morris T, Armstrong J, Wirth MP; Casodex Early Prostate Cancer Trialists' Group. Bicalutamide 150 mg plus standard care vs standard care alone for early prostate cancer. BJU Int. 2006 Feb;97(2):247-54. doi: 10.1111/j.1464-410X.2005.06051.x. PMID 16430622
- [Background] Ramirez AG, Trapido EJ. Advancing the Science of Cancer in Latinos. 2022 Nov 15. In: Ramirez AG, Trapido EJ, editors. Advancing the Science of Cancer in Latinos: Building Collaboration for Action [Internet]. Cham (CH): Springer; 2023. Chapter 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK595808/ PMID 37816115
- [Background] Potosky AL, Davis WW, Hoffman RM, Stanford JL, Stephenson RA, Penson DF, Harlan LC. Five-year outcomes after prostatectomy or radiotherapy for prostate cancer: the prostate cancer outcomes study. J Natl Cancer Inst. 2004 Sep 15;96(18):1358-67. doi: 10.1093/jnci/djh259. PMID 15367568

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT07339943/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT07339943/ICF_001.pdf